CLINICAL TRIAL: NCT02664454
Title: Compared Efficacy of Nurse-led and GP-led Geriatric Assessment in PrImary Care: A Pragmatic Three-arm Cluster Randomized Controlled Trial
Brief Title: Compared Efficacy of Nurse-led and GP-led Geriatric Assessment in PrImary Care
Acronym: CEPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K140707
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multimorbidity; Geriatric Assessment
Keywords: Elderly; Health care organization; Primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Systematic nurse-led GA (Experimental): Interactive educational seminar for GPs and nurses, and focused on geriatric assessment in primary care combined with Systematic nurse-led GA and dedicated hotline for GPs seeking geriatric advice
  Interventions: Other: health care organization
- GP-led GA on a case-by-case basis, as decided by the GP (Experimental): Interactive educational seminar for GPs, and focused on Geriatric assessment in primary care combined with a GP-led GA on a case-by-case basis, as decided by the GP, and a dedicated hotline for GPs seeking geriatric advice
  Interventions: Other: health care organization
- No intervention (No Intervention): No educational seminar Usual care

INTERVENTIONS:
Other: health care organization — Nurse-led or GP-led Geriatric assessment combined with an educational seminar focused on GA and personalized care-plan as well as a dedicated hotline for general practitioners seeking a geriatric advice
  Interactive educational seminar Primary care
  Other Names: Nurse-led or GP-led Geriatric assessment combined with an educational seminar
  Arms: GP-led GA on a case-by-case basis, as decided by the GP; Systematic nurse-led GA

SUMMARY:
Older patients account for around 10% of the population, of which 57% have a long-term illness, and 33% were admitted in the past year.

Geriatric assessment (GA) is a multidimensional assessment of general health status that can help identifying deficiencies and followed by a personalized care plan.

Assessment and management of elderly patients is a daily concern for the general practitioner (GP) but conflicting results have been reported so far relating to the clinical impact of GA when applied in the primary care setting.

This study protocol aims to assess the effect on morbi-mortality of a complex intervention in patients aged ≥70 years with chronic conditions in primary care. It aims to demonstrate that a GA adapted to primary care, followed by a personalized care plan and combined with successful interprofessional collaboration can improve clinically relevant outcomes in elderly patients with chronic conditions such as one-year overall mortality, unplanned hospital admission, emergency visits, or institutionalization.

The CEPIA study will also help addressing the issue of whether an improved benefit could be achieved from a systematic nurse-led or a case-by-case GP-led GA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged≥70 years with a long-term illness scheme or hospital admission the past 3 months
* Visiting their preferred general practioner (GP) or another GP in the same practice
* patient oral non opposition

Exclusion Criteria:

* Patient who does not speak French
* Severe disease with a life expectancy <12 months
* Institutionalized patients
* Patient insured under the French national health insurance system

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 750 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Primary composite endpoint combined with: - Percentage of all-cause mortality - Percentage of Unplanned hospital admission - Percentage of Emergency visits. - Percentage of Institutionalization | At 12 months

SECONDARY OUTCOMES:
Percentage of all-cause mortality | At 12 months
Percentage of Unplanned hospital admission | At 12 months
Percentage of Emergency visits | At 12 months
Percentage of Institutionalization | At 12 months
Quality of life (Duke profile score) | At Day 0 and 12 months
Autonomy by KATZ ALD score | At Day 0 and 12 months
Number of medication prescription (polypharmacy) | Up to 12 months
Percentage of Geriatric assessment performed | Up to 12 months
Percentage of personalized care plan performed | Up to 12 months
Percentage of geriatric phone advices requested by GPs | Up to 12 months
Percentage of health care actions planned | Up to 12 months
Percentage of satisfied general practitioner with the intervention | 27months after the beginning of the study
  self-assessment
Satisfaction of general practitioners and nurses after completion of intervention | 12 months after the beginning of the study
  interview of general practionners and nurses by independant investigator

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Ferrat, MCU-MG, Principal Investigator — Université Paris Est (UPEC), IMRB, A-TVB DHU, CEpiA EA 7376 (Clinical Epidemiology and Ageing Unit)
Locations (1):
- Faculté de Médecine, Université Paris Est Créteil (UPEC), Créteil, France

REFERENCES:
- [Result] Bouman A, van Rossum E, Nelemans P, Kempen GI, Knipschild P. Effects of intensive home visiting programs for older people with poor health status: a systematic review. BMC Health Serv Res. 2008 Apr 3;8:74. doi: 10.1186/1472-6963-8-74. PMID 18387184
- [Result] Kuo HK, Scandrett KG, Dave J, Mitchell SL. The influence of outpatient comprehensive geriatric assessment on survival: a meta-analysis. Arch Gerontol Geriatr. 2004 Nov-Dec;39(3):245-54. doi: 10.1016/j.archger.2004.03.009. PMID 15381343
- [Result] Stuck AE, Siu AL, Wieland GD, Adams J, Rubenstein LZ. Comprehensive geriatric assessment: a meta-analysis of controlled trials. Lancet. 1993 Oct 23;342(8878):1032-6. doi: 10.1016/0140-6736(93)92884-v. PMID 8105269
- [Result] Stuck AE, Egger M, Hammer A, Minder CE, Beck JC. Home visits to prevent nursing home admission and functional decline in elderly people: systematic review and meta-regression analysis. JAMA. 2002 Feb 27;287(8):1022-8. doi: 10.1001/jama.287.8.1022. PMID 11866651
- [Result] Frese T, Deutsch T, Keyser M, Sandholzer H. In-home preventive comprehensive geriatric assessment (CGA) reduces mortality--a randomized controlled trial. Arch Gerontol Geriatr. 2012 Nov-Dec;55(3):639-44. doi: 10.1016/j.archger.2012.06.012. Epub 2012 Jul 11. PMID 22790107
- [Result] Ellis G, Whitehead MA, O'Neill D, Langhorne P, Robinson D. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD006211. doi: 10.1002/14651858.CD006211.pub2. PMID 21735403
- [Result] Li CM, Chen CY, Li CY, Wang WD, Wu SC. The effectiveness of a comprehensive geriatric assessment intervention program for frailty in community-dwelling older people: a randomized, controlled trial. Arch Gerontol Geriatr. 2010 Feb;50 Suppl 1:S39-42. doi: 10.1016/S0167-4943(10)70011-X. PMID 20171455
- [Derived] Orcel V, Ferrat E, Moscova L, Vigneron L, Michau B, Cittee J, Adeline F, Audureau E, Hagege M. Barriers to and facilitators of comprehensive geriatric assessment in primary care in France: a qualitative study exploring physicians' and nurses' experiences. BMC Prim Care. 2025 Dec 30;26(1):414. doi: 10.1186/s12875-025-03085-5. PMID 41469541
- [Derived] Orcel V, Banh L, Bastuji-Garin S, Renard V, Boutin E, Gouja A, Caillet P, Paillaud E, Audureau E, Ferrat E. Effectiveness of comprehensive geriatric assessment adapted to primary care when provided by a nurse or a general practitioner: the CEpiA cluster-randomised trial. BMC Med. 2024 Sep 27;22(1):414. doi: 10.1186/s12916-024-03613-7. PMID 39334117
- [Derived] Ferrat E, Bastuji-Garin S, Paillaud E, Caillet P, Clerc P, Moscova L, Gouja A, Renard V, Attali C, Breton JL, Audureau E. Efficacy of nurse-led and general practitioner-led comprehensive geriatric assessment in primary care: protocol of a pragmatic three-arm cluster randomised controlled trial (CEpiA study). BMJ Open. 2018 Apr 12;8(4):e020597. doi: 10.1136/bmjopen-2017-020597. PMID 29654038